CLINICAL TRIAL: NCT02684526
Title: Is Eovist Suitable for Arterial-Phase MR Imaging of Liver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hero Hussain, MD, Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: HUM00038856
Record Dates: First submitted 2013-03-14; First posted 2016-02-18 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-10

CONDITIONS: Liver Disease
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eovist Contrast agent (Active Comparator): To determine if Eovist contrast agent induces a transient abnormal sensation at first pass, which prevents patients from holding their breath at end of arterial phase liver MRI scans.
  Interventions: Procedure: Eovist Contrast
- Non Eovist Contrast agents (Active Comparator): To determine if using non-Eovist contrast agents produce the same abnormal sensation at first pass, which prevents patients from holding their breath at end of arterial phase liver MRI scans. Determine if this event is exclusive to Eovist contrast.
  Interventions: Procedure: Non Eovist Contrast

INTERVENTIONS:
Procedure: Eovist Contrast — Subjects will undergo an MRI (magnetic resonance imaging) scan using the Eovist contrast agent. This MRI scan takes approximately 45minutes to 1 hour to complete.
  Arms: Eovist Contrast agent
Procedure: Non Eovist Contrast — Subjects will undergo an MRI (magnetic resonance imaging) scan using a contrast agent other than Eovist. This MRI scan takes approximately 45minutes to 1 hour to complete.
  Arms: Non Eovist Contrast agents

SUMMARY:
To examine the quality of liver images produced when the contrast agent Eovist is used during MRI.

DETAILED DESCRIPTION:
Researchers will review data from the Eovist MRI and compare the scan with previous MRI exams the patient had with the same or other contrast agents.

To determine the efficacy of Eovist contrast agent in producing MRI images of the liver. We will monitor patients for any unusual symptoms (adverse events) when the contrast is given.

Patients are asked to hold their breath during an MRI scan. Eovist may interfere with the "breath hold" which could result in more breathing artifacts (based on a qualitative scale) on arterial images when the patients are given Eovist vs. other contrast agents.

ELIGIBILITY:
Inclusion Criteria:

1. You have had a scheduled MRI(magnetic resonance imaging) scan using the contrast agent EOVIST.
2. Male and females 21 years of age or older.

Exclusion Criteria:

1. Does not have a contraindication for MRI (e.g. cardiac pacemaker, ferromagnetic or metallic implants).
2. Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2011-12; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Scanning artifacts on MRI with Eovist | 5 years
  To qualitatively assess and score MRI images during unenhanced and contrast-enhanced motion-sensitive sequences for breathing artifacts when Eovist contrast is used versus other contrast agents. Eovist enhanced MRI scans will be compared to previous MRI scans performed with other contrast agents on the same patient that included breath holding sequences. Breathing artifacts on both scans will be evaluated using a respiratory motion score between 1 and 5.

SECONDARY OUTCOMES:
Adverse events (including dyspnea) | 30 min
  Number of patients complaining of adverse events after MRI contrast administration.

CONTACTS AND LOCATIONS:
Overall Officials: Hero Hussain, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No